CLINICAL TRIAL: NCT02587026
Title: Collection of Specimens and Clinical Data to Create a Biorepository for Precision Genomics
Brief Title: Biorepository for Precision Genomics
Status: Terminated | Type: Observational
Why Stopped: Study team has decided to close enrollment, and all subjects are being rolled into a different clinical trial: Total Cancer Care
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Bryan Schneider, Clinical Pharmacy Specialist, Indiana University
Other Study IDs: IUSCC-0534
Record Dates: First submitted 2015-10-08; First posted 2015-10-27 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Neoplasms
Keywords: Biorepository; Precision Genomics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Biospecimen Retention: Samples With DNA — Prospective blood and tumor tissue samples will be collected. Retrospective review of patient charts for clinical information will also be done.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood sample collection
Other: Tumor tissue sample collection

SUMMARY:
This is a tissue collection protocol to create an annotated biorepository to support future basic and translational research. The study protocol and consent will request patient permission to allow their specimens to be stored for future use in other laboratory/correlative studies without requiring a separate new consent at a future date. It will include also a retrospective review of all patients who have been seen or treated by the Precision Genomics Clinic (waiver of consent requested). No specific research studies/aims are included directly in this proposal. Use of the samples, data, and other resources (cell lines, etc.) created within this protocol will require review/approval by the majority of the Precision Genomics Investigators and appropriate IRB approval.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Patients must have histologically or cytologically confirmed malignancy or related disorder. This includes patients with active disease as well as those in remission.
4. One of the following tissue collection situations

   * Group 1: Patients having tissue collection for clinical reasons who are willing to have additional specimens taken for research (biopsy may be done under local anesthesia, intravenous conscious sedation, or general anesthesia, as clinically indicated)
   * Group 2: Patients willing to undergo tissue collection for the purpose of research only (biopsy may be done under local anesthesia or intravenous conscious sedation per the judgment of the treating physician). This may include collection of additional samples from patients undergoing a study-specific research biopsy/procedure. Patients in group 2 may not undergo general anesthesia as part of this protocol.
   * Group 3: Patients having tissue collection for clinical reasons who are willing to have excess tissue (i.e., tissue that would have otherwise been discarded) banked for research (biopsy may be done under local anesthesia, intravenous conscious sedation, or general anesthesia, as clinically indicated).
5. Willingness to undergo phlebotomy for research blood samples Additional Criteria for Patients in Groups 1 and 2
6. PT and PTT levels < 1.2 x the institutional ULN (PT, PTT not required for skin biopsies)
7. Not receiving therapeutic anticoagulation
8. Platelets ≥ 100 x 109/L

Exclusion Criteria:

1. Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety.
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
3. History of serious or life-threatening allergic reaction to local anesthetics (i.e. lidocaine, xylocaine)
4. Any other condition, which in the opinion of the patient's treating oncologist or the physician performing the biopsy procedure, would make participation in this protocol unreasonably hazardous for the patient.

   Additional Criteria for Patients in Group 1 and 2
5. Pregnant women are excluded from Groups 1 and 2 because there may be an increased risk to both mother and fetus in the setting of conscious sedation, which is required for biopsies of certain anatomic sites (e.g. liver, lung, bone). Also, ionizing radiation from CT-guided biopsies may pose a risk to the unborn fetus.
6. Patients in Groups 1 and 2 may not have active cardiac disease, defined as:

   * History of uncontrolled or symptomatic angina
   * History of arrhythmias requiring medications, or clinically significant
   * Myocardial infarction < 6 months from study entry
   * Uncontrolled or symptomatic congestive heart failure
   * Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
7. Patients in group 1 and 2 receiving bevacizumab or other angiogenesis inhibitors (or less than 6 weeks from last dose of an angiogenesis inhibitor) should not undergo a research core liver biopsy on this protocol because of the concern for the possibility of increased bleeding risk. Patients may undergo a research fine needle aspiration (FNA) of the liver as an alternative. Patients may also undergo core research biopsies of other sites, up to the discretion of the treating physician, but physicians should take the potential increased bleeding and/or delayed wound healing issues into consideration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attend the Precision Genomics Clinic at Indiana University Health may elect to participate in this tissue and blood collection protocol.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Biorepository for precision genomics | From time of patient consent (day 1) to time of sample collection (which can occur on day 1-day 35)
  Blood and tissue sample collection for use in future basic and translational research studies

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Schneider, MD, Principal Investigator — Vera Bradley Professor of Oncology, Professor of Medicine, Professor of Medical & Molecular Genetics
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Ball Memorial, Muncie, Indiana